CLINICAL TRIAL: NCT02609113
Title: A Double Blinded, Prospective, Randomized Trial of Static Magnetic Therapy for Carpal Tunnel Syndrome (CTS)
Brief Title: Static Magnetic Therapy for Carpal Tunnel Syndrome
Acronym: ATTRACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTS-MAG-22
Record Dates: First submitted 2015-11-13; First posted 2015-11-20 (Estimated); Results first posted 2018-01-16 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Strong Magnetic Wristband (Active Comparator): Magnetic wristband of 1,795 Gauss strength
  Interventions: Device: Strong Magnetic Wristband
- Weaker Magnetic Wristband (Placebo Comparator): Magnetic wristband of 5 Gauss strength.
  Interventions: Device: Weaker Magnetic Wristband

INTERVENTIONS:
Device: Strong Magnetic Wristband
  Arms: Strong Magnetic Wristband
Device: Weaker Magnetic Wristband
  Arms: Weaker Magnetic Wristband

SUMMARY:
The purpose of this research study is to investigate if magnet therapy is effective as an alternative therapy for CTS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild to moderate Carpal Tunnel Syndrome by history, clinical exam and Electromyography (EMG) study.
* ≥ 18 years

Exclusion Criteria:

* Current use of magnets as therapy for Carpal Tunnel Syndrome
* Known allergy to silicone
* Unwillingness to wear wristband for 6 weeks
* Patients who have devices that may be affected by exposure to magnets such as vagal nerve stimulator, pacemaker or insulin pump.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-08; Primary Completion 2016-10-21 (Actual); Study Completion 2016-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Baute, MD, Principal Investigator — Wake ForestUBMC
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Strong Magnetic Wristband: Magnetic wristband of 1,795 Gauss strength
  Strong Magnetic Wristband
- Weaker Magnetic Wristband: Magnetic wristband of 5 Gauss strength.
  Weaker Magnetic Wristband
Period: Overall Study
Arm/Group | Strong Magnetic Wristband | Weaker Magnetic Wristband
Started | 11 | 11
Completed | 9 | 9
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Strong Magnetic Wristband | Weaker Magnetic Wristband | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Median (Standard Deviation); unit: years] | 46 (9.60) | 52 (6.12) | 48.7 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 0 | 3 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Boston Carpal Tunnel Questionnaire (BCTQ) Score at 6 Weeks
Description: Patient reported outcome measure of symptom severity and functional status. Is made of the Symptom severity scale (11 items) score 1 to 5 where lower numbers denotes better outcomes; and the Functional status scale (8 items) score 1 to 5 where lower numbers denotes better outcomes. Total score 1- 95 where lower numbers denotes better outcomes.
Time Frame: Baseline and 6 weeks
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Strong Magnetic Wristband | Weaker Magnetic Wristband
Number analyzed (Participants) | 9 | 9
units on a scale | 48.6 (6.6) | 45.4 (4.5)

2. Secondary Outcome: Change in Echogenicity (Hyper or Hypo) on the Median Nerve Ultrasound at 6 Weeks
Description: Ultrasound to assess the anatomy of the median nerve
Time Frame: Baseline and 6 weeks
Population: The Median Nerve Echogenicity (% hypoechoic) was the same at 89%.
Measure: Number; unit: percentage of hypoechoic
Arm/Group | Strong Magnetic Wristband | Weaker Magnetic Wristband
Number analyzed (Participants) | 9 | 9
percentage of hypoechoic | 89 | 89

3. Secondary Outcome: Change in Cross-sectional Area as Measured in mm2 on Median Nerve Ultrasound at 6 Weeks
Description: Ultrasound to assess the anatomy of the median nerve
Time Frame: Baseline and 6 weeks
Measure: Median (Standard Deviation); unit: mm^2
Arm/Group | Strong Magnetic Wristband | Weaker Magnetic Wristband
Number analyzed (Participants) | 9 | 9
mm^2 | 11.6 (2.8) | 14.2 (3.5)

4. Secondary Outcome: Change in Vascularity (Normal or Abnormal) as Measured on Median Nerve Ultrasound at 6 Weeks
Description: Ultrasound to assess the anatomy of the median nerve
Time Frame: Baseline and 6 weeks
Measure: Number; unit: percentage of Abnormal
Arm/Group | Strong Magnetic Wristband | Weaker Magnetic Wristband
Number analyzed (Participants) | 9 | 9
percentage of Abnormal | 33 | 33

ADVERSE EVENTS:
Time Frame: Baseline to 6 weeks
Arm/Group | Strong Magnetic Wristband | Weaker Magnetic Wristband
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

LIMITATIONS AND CAVEATS:
Limitations of the study that could contribute to the lack of measurable change include a short duration, small sample size, and inefficacy of magnet therapy in relation to neurodiagnostic measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No